CLINICAL TRIAL: NCT05365438
Title: Effect of Atorvastatin and Omega 3 Combination Therapy on Carotid Atherosclerosis Estimated by 3D Ultrasound in Patients With Type 2 Diabetes and Combined Dyslipidemia
Brief Title: Atmeg (Atorvastatin and Omega-3 Combination) and Carotid Atherosclerosis in Patients With Type 2 Diabetes and Combined Dyslipidemia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Korea United Pharm. Inc. (Industry)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-2111-720-004
Record Dates: First submitted 2022-04-27; First posted 2022-05-09 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Dyslipidemias; Atherosclerosis; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Dyslipidemias; Atherosclerosis; Diabetes Mellitus, Type 2 | interventions — liptruzet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Atmeg with Omethyl Cutielet (Experimental): Atmeg: 2 capsules daily (1 capsule containes atorvastatin 10 mg and Omega-3 1000 mg) Omethyl Cutielet: Omega-3 2000mg (920mg as EPA ethyl ester, 760mg as DHA ethyl ester) once daily
  Interventions: Drug: Omega 3-Atorvastatin
- Atmeg (Active Comparator): Atmeg: 2 capsules daily (1 capsule containes atorvastatin 10 mg and Omega-3 1000 mg)
  Interventions: Drug: Omega 3-Atorvastatin
- ezetimibe/atorvastatin 10/20 (Active Comparator): 1 tablet once daily (atorvastatin 20mg with ezetimibe 10mg)
  Interventions: Drug: Atorvastatin-Ezetimibe

INTERVENTIONS:
Drug: Omega 3-Atorvastatin — Atmeg 2 capsules with 1 pack of Omethyl cutielet
  Other Names: Atmeg-Omethyl cutielet
  Arms: Atmeg with Omethyl Cutielet
Drug: Omega 3-Atorvastatin — Atmeg 2 capsules
  Other Names: Atmeg
  Arms: Atmeg
Drug: Atorvastatin-Ezetimibe — ezetimibe/atorvastatin 10/20 mg
  Arms: ezetimibe/atorvastatin 10/20

SUMMARY:
This is a randomized controlled study to assess the effect of atorvastatin and omega 3 combination therapy compared with atorvastatin and ezetimibe combination therapy in Korean T2DM patients with asymptomatic atherosclerosis.

DETAILED DESCRIPTION:
In patients with type 2 diabetes with atherosclerotic combined dyslipidemia, the effect of atorvastatin and omega 3 combination on the progression of carotid intima media thickness and carotid artery plaque will be evaluated by 3D carotid ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes under treatment with HbA1c 6.0-10.0% at screening visit
* Male or female of 20 years or over
* Mixed dyslipidemia under moderate-intensity statin: triglyceride ≥200 mg/dL, HDL-cholesterol ≤50 mg/dL, LDL-cholesterol ≥100 mg/dL

  * moderate-intensity statin: atorvastatin 10-20mg, rosuvastatin 5mg, simvastatin 20-40mg, pravastatin 40-80mg, lovastatin 40mg, fluvastatin XL 80mg, fluvastatin 40mg bid, pitavastatin 2-4mg
* Identified carotid artery plaque: carotid intima-media thickness (cIMT) ≥ 1.0 mm
* Asymptomatic patients without history of angina, myocardial infarction, or cerebral infarction
* Creatinine ≤1.8 mg/dL

Exclusion Criteria:

* Dyslipidemia which requires other therapy: triglyceride ≥500 mg/dL or LDL-cholesterol ≥190 mg/dL
* Uncontrolled hypertension: SBP >180 mmHg or DBP >110 mmHg
* Severe renal dysfunction: eGFR <30 mL/min/1.73m2
* AST/ALT >120/120 or chronic liver disease
* Pregnant or childbearing woman who does not have enough contraception
* Changes of medication related to chronic diseases (diabetes, hypertension, dyslipidemia, etc.) within 3 months
* Usage of dyslipidemia therapy other than statin

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Carotid intima media thickness | 24 weeks
  maximum carotid IMT (mm)

SECONDARY OUTCOMES:
Area of carotid artery plaque | 24 weeks
  measured by ultrasound
Plaque characteristics Plaque characteristics Plaque characteristics Plaque characteristics | 24 weeks
  changes of non-calcified plaque volume (mm3)
Glucose homeostasis | 24 weeks
  changes of HbA1c (%)
Lipid metabolism | 24 weeks
  TG concentration, HDL-cholesterol concentration
Bioelectrical Impedance Analysis | 24 weeks
  Body composition of fat mass (kg)
Proteinuria | 24 weeks
  albumin-to-creatinine ratio (mg/g)
Changes of gut microbiota | 24 weeks
  measured by 16S rRNA or metagenome sequencing, comparing the composition or each phylum/genus/species

CONTACTS AND LOCATIONS:
Locations (1):
- SNUBH, Seongnam-si, Gyeonggi-do, South Korea